CLINICAL TRIAL: NCT04966663
Title: From Liquid Biopsy to Cure: Using ctDNA Detection of Minimal Residual Disease to Identify Patients for Curative Therapy After Lung Cancer Resection
Brief Title: Using ctDNA to Determine Therapies for Lung Cancer
Acronym: ctDNA Lung RCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ctDNA Lung RCT
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer; Complete Surgical Resection; Circulating Tumor DNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Pemetrexed; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant chemo-immunotherapy therapy (Experimental): All participants will have blood taken for ctDNA testing.
  A cycle is 21 days. Pemetrexed (for participants with non-squamous non-small cell lung cancer), intravenously (by vein) on Day 1 of Cycles 1-4, OR gemcitabine (for all other participants) on Days 1 and 8 of Cycles 1-4.
  Cisplatin*, intravenously (by vein) on Day 1 of Cycles 1-4 Nivolumab, intravenously (by vein) on Day 1 of Cycles 1-4
  *If cisplatin is not tolerated, carboplatin may be given instead
  Interventions: Drug: Nivolumab; Drug: Pemetrexed; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin; Procedure: ctDNA blood test
- Observation (Other): All participants will have blood taken for ctDNA testing.
  Participants will be followed as per standard of care every 3 months.
  Interventions: Procedure: ctDNA blood test

INTERVENTIONS:
Drug: Nivolumab — Antineoplastic agent
  Other Names: Opdivo; ONO-4538; BMS-936558; MDX1106
  Arms: Adjuvant chemo-immunotherapy therapy
Drug: Pemetrexed — Antineoplastic agent
  Other Names: Alimta; Pemfexy
  Arms: Adjuvant chemo-immunotherapy therapy
Drug: Gemcitabine — Antineoplastic agent
  Other Names: Gemzar; 2'; 2'-difluoro 2'deoxycytidine; dFdC
  Arms: Adjuvant chemo-immunotherapy therapy
Drug: Cisplatin — Antineoplastic agent
  Other Names: Cisplatinum; platamin; neoplatin; cismaplat; cis-diamminedichloroplatinum(II) (CDDP); Platinol; Platinol-AQ
  Arms: Adjuvant chemo-immunotherapy therapy
Drug: Carboplatin — Antineoplastic agent
  Other Names: Paraplatin; Paraplatin-AQ; CBDCA; JM8; NSC 241240; Paraplatin NovaPlus
  Arms: Adjuvant chemo-immunotherapy therapy
Procedure: ctDNA blood test — Blood will be collected for ctDNA testing

SUMMARY:
This is a study to look at whether the presence of circulating tumour DNA (ctDNA) in the blood can help to predict whether giving adjuvant treatment after surgery can decrease the chance of the cancer coming back in people with lung cancer.

DETAILED DESCRIPTION:
For people who have early stage non-small cell lung cancer (NSCLC), the usual treatment is surgery. For many people, surgery is enough to get rid of all the cancer. However, for some people, there may be a little bit of cancer remaining. If there is some cancer left over, it may lead to the cancer regrowing. This is called relapse.

Many cancers shed little bits of their DNA (deoxyribonucleic acid, molecules that contain instructions for how cells develop and function) into the bloodstream. A blood test can be used to test for the amount of circulating tumour DNA (ctDNA). Some studies have shown that the presence of ctDNA in the blood may predict cancer recurrence.

The purpose of this research study is to see if adjuvant treatment (additional treatment given after primary treatment) can help decrease the risk of the cancer recurring in people with lung cancer who have ctDNA detected in their blood after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of screening
2. Written informed consent obtained from the subject prior to performing any protocol-related procedures
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Weight ≥ 35 kg
5. Must have a life expectancy of at least 24 months
6. Complete surgical resection of T1-2N0M0 NSCLC or T3/T4 multifocal NSCLC
7. Any pathologic subtype of NSCLC is eligible, including adenocarcinoma and squamous carcinoma. Patients with targetable genomic alterations without approved or available targeted adjuvant therapy options are eligible
8. Patients with detectable plasma ctDNA before or after complete surgical resection are eligible (RaDaR TM assay, Inivata Morrisville, North Carolina, USA).
9. No prior chemotherapy or radiotherapy is allowed for the current diagnosis of resected NSCLC.
10. Adequate organ and marrow function as defined in Table 4 (3.1.1)
11. Females of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception from screening to 180 days after the final dose of study treatment. A serum pregnancy test within 72 hours prior to the initiation of therapy will be required for women of childbearing potential. It is strongly recommended for the male partner of a female subject to also use male condom plus spermicide throughout this period
12. Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use a male condom with spermicide from screening to 180 days after receipt of the final dose of study treatment. It is strongly recommended for the female partner of a male subject to also use a highly effective method of contraception throughout this period. In addition, male subjects must refrain from sperm donation while on study and for 180 days after the final dose of study treatment.

4.1.2 Exclusion Criteria

1. Participants that should receive adjuvant chemotherapy per standard of care (resected N1 or N2 disease, primary tumour >=4 cm).
2. Receipt of any conventional or investigational anticancer therapy within 21 days or radiotherapy within 14 days prior to the scheduled first dose of study treatment;
3. Prior receipt of any immune-mediated anti-cancer therapy including, but not limited to, anti-CTLA-4, anti-PD-1, anti-PD-L1 antibodies including nivolumab and agents targeting CD73, CD39, or adenosine receptors;
4. Incomplete surgical resection;
5. Concurrent enrolment in another therapeutic clinical study of systemic anti-cancer treatment. Enrolment in observational or supportive studies will be allowed;
6. Subjects with a recent history of myocardial infarction, congestive heart failure ≥ Class 3 based on New York Heart Association Functional Classification or stroke within the past 3 months prior to the scheduled first dose of study treatment;
7. Active autoimmune disorders within the past 3 years prior to the scheduled first dose of study treatment. The following are exceptions to this criterion:

   1. Subjects with vitiligo or alopecia.
   2. Subjects with hypothyroidism (e.g., following Hashimoto syndrome) not requiring systemic treatment or stable on hormone replacement.
   3. Subjects with psoriasis not requiring systemic treatment.
   4. Any chronic skin condition that does not require systemic therapy.
   5. Subjects with celiac disease controlled by diet alone;
8. Have known uncontrolled human immunodeficiency virus (HIV)-1/2 infection.

   • Participants with HIV (known HIV 1/2 antibodies positive) are allowed if all of the following conditions are met: CD4+ T-cell counts ≥350 cells/uL; no opportunistic infection within the past 12 months; on established anti-retroviral therapy for at least 4 weeks; and an HIV viral load less than 400 copies/mL.
9. History of primary immunodeficiency, solid organ transplantation, or active tuberculosis (by clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice). In settings where there is clinical or radiographic evidence of tuberculosis, active disease must be excluded prior to enrolment. Subjects who have had adequately treated tuberculosis may be enrolled upon discussion with the coordinating Principal Investigator.
10. Other invasive malignancy within 2 years. Non-invasive malignancies (i.e., cervical carcinoma in situ, in situ prostate cancer, non-melanomatous carcinoma of the skin, ductal carcinoma in situ of the breast that has been surgically cured) are permitted.
11. Known allergy or hypersensitivity to investigational product formulations.
12. History of more than one event of infusion related reactions (IRR) requiring permanent discontinuation of IV drug treatment.
13. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring antibiotic therapy, uncontrolled hypertension, bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs, or compromise the ability of the subject to give written informed consent.
14. Current or prior use of immunosuppressive medication within 14 days prior to the scheduled first dose of study treatment. The following are exceptions to this criterion:

    1. Intranasal, topical, inhaled corticosteroids or local steroid injections (e.g., intra articular injection).
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent.
    3. Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication).
15. Receipt of live, attenuated vaccine within 30 days prior to the scheduled first dose of study treatment (Note: Subjects, if enrolled, should not receive live vaccine during the study and 180 days after the last dose of study treatment). Vaccination with an inactivated vaccine is permitted at any time.
16. Major surgery (as defined by the investigator) within 28 days prior to the scheduled first dose of study treatment or still recovering from prior surgery. Local procedures (e.g., placement of a systemic port, core needle biopsy, etc) are allowed without needing to wait for the 28-day recovery period.
17. Females who are pregnant, lactating, or intend to become pregnant during their participation in the study.
18. Subjects who are involuntarily incarcerated or are unable to willingly provide consent or are unable to comply with the protocol procedures.

    Any condition that, in the opinion of the investigator, would interfere with safe administration or evaluation of the investigational products or interpretation of subject safety or study results
19. Any condition that, in the opinion of the investigator, would interfere with safe administration or evaluation of the investigational products or interpretation of subject safety or study results.
20. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Nivolumab or other agents used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival | 2 years
  To demonstrate the impact of intensified adjuvant therapy on relapse-free survival (RFS) in patients at high risk of relapse post-resection identified by pre- or post-operative detectable ctDNA plasma levels in patients with resected T1-T4 (T3-4 multifocal only) N0M0 NSCLC.

SECONDARY OUTCOMES:
Rate of ctDNA clearance | 12 weeks
  To estimate and compare the ctDNA detection rates at 12 weeks post-randomization in those receiving adjuvant chemo-immunotherapy versus observation.
Overall survival | 3 years
  To compare overall survival (OS) of patients receiving adjuvant chemo-immunotherapy versus observation.
Number of adverse events | 3 years
  To determine safety and tolerability of adjuvant chemo-immunotherapy with the combination of nivolumab with cisplatin and pemetrexed or nivolumab with cisplatin and gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Leighl, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada